CLINICAL TRIAL: NCT02469935
Title: Accuracy of Surgeon-performed Ultrasound in Detecting Gallstones - a Validation Study
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Camilla Gustafsson, PhD student, Karolinska Institutet
Other Study IDs: 2011/1025-31/1
Record Dates: First submitted 2015-06-03; First posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Gallstones
Keywords: Validation; Surgeon-performed ultrasound; Gallstones
MeSH Terms: conditions — Gallstones | interventions — High-Energy Shock Waves

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ultrasound — surgeon-performed ultrasound

SUMMARY:
Aims: To prospectively investigate the accuracy of surgeon-performed ultrasound for the detection of gallstones.

Methods: 179 adult patients, with an acute or elective referral for an abdominal ultrasound examination, were examined with a right upper quadrant ultrasound scan by a radiologist as well as surgeon. The surgeons had undergone a four-week long education in ultrasound before participating in the study. Ultrasound findings of the surgeon were compared to those of the radiologist, using radiologist-performed ultrasound as reference standard.

DETAILED DESCRIPTION:
Enrolment of patients:

Three hundred patients, with an acute or elective referral to the radiology department at Stockholm South General Hospital, Sweden, for any diagnostic abdominal US examination, including both patients admitted to in-hospital care and out-patients, were prospectively enrolled between October 2011 and November 2012. Eligible patients were identified in the radiology department by a study surgeon and informed consent was obtained. Six US educated surgeons participated in the enrolment of patients. Exclusion criteria were age <18 years or inability to communicate with the examiner. Referrals concerning metastases of the liver or contrast-enhanced examinations were considered not suitable for the study and were also excluded. The surgeons examined patients consecutively if time was available, but mostly they didn't have time to examine every patient referred per day, hence a certain prioritisation between referrals was done.

Data collection:

Enrolled patients received one US examination by the study surgeon as well as the standard US examination by the on-duty radiologist. In a majority of cases the two examinations were performed consecutively and the time interval between the surgeon-performed US and radiologist-performed US never exceeded 24 hours. The surgeon's examination took place either before or right after the radiologist's examination. The examining surgeon and radiologist were blinded to each other's findings. The surgeon's US examination followed a standardised protocol, which included a full abdominal scan, regardless of the nature of the referral. The presence of gallstones was marked as a 'yes' (positive finding, regardless of number or size) or 'no' (negative finding) by the surgeon. In cases where a full abdominal scan could not be performed, due to urgent patient management, a focused examination based on the referral as well as a right upper quadrant (RUQ) scan was advised. The on-duty radiologist performed a standard care US focusing on the individual referrals. The radiologist's statement was collected from the patient's medical record and transferred to the study protocol by a separate radiologist, who was also blinded to the surgeon's examination. Among the radiologists the major part of the scans was done by US specialised radiologists with several years of training (56% US specialists, 73% specialists in radiology).

The surgeons used a portable US machine of the model LOGIQ e with a convex (1.6-4.6 MHz) or linear (5-13 MHz) transducer, GE Healthcare, WuXi, China. All scans were saved on a separate hard drive, which was kept together with the study protocol. The radiologists used Philips iU22 with a convex C5-1 or a linear L12-5 transducer.

US training of surgeons participating in the study:

Six study surgeons, five in the final years of their specialist training and one specialist in surgery, with limited or no previous US training, attended a one-week course, comprising US physics, technique, anatomy and hands-on training, led by specialists in US. After attending the course the surgeons received three weeks of training in the radiology department under the guidance of an US specialist. The surgeons were expected to perform a minimum of 50 supervised scans, which was obtained in all cases but one. The training focused on detecting gallbladder stones, widened bile ducts, thickened wall of the gallbladder, lesions in the liver parenchyma, hydronephrosis, abdominal aortic aneurysms, free abdominal fluid and appendicitis. After the training was completed, each surgeon spent a minimum of two weeks enrolling and scanning patients during office hours in the hospital's radiology department.

Ethics:

The patients received oral and written information from the study surgeon and were included after informed consent. The study was approved by the Ethical Review Board, at Karolinska Institutet, Stockholm, Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the radiology department for an abdominal ultrasound
* Age > 18 years

Exclusion Criteria:

* Inability to communicate with the examiner
* Referral for intervention
* Metastasis screening
* Referrals concerning contrast enhanced examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the radiology department for an abdominal ultrasound.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Accuracy of surgeon-performed ultrasound | 13 months
  Compared to radiologist-performed ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Anders Sonden, MD. PhD, Principal Investigator — Karolinska Institutet Södersjukhuset
Locations (1):
- Karolinska Institutet Södersjukhuset (South General Hospital), Stockholm, Stockholm County, Sweden

REFERENCES:
- [Result] Powers RD, Guertler AT. Abdominal pain in the ED: stability and change over 20 years. Am J Emerg Med. 1995 May;13(3):301-3. doi: 10.1016/0735-6757(95)90204-X. PMID 7755822
- [Result] Cooperberg PL, Burhenne HJ. Real-time ultrasonography. Diagnostic technique of choice in calculous gallbladder disease. N Engl J Med. 1980 Jun 5;302(23):1277-9. doi: 10.1056/NEJM198006053022303. PMID 7366693
- [Result] Kell MR, Aherne NJ, Coffey C, Power CP, Kirwan WO, Redmond HP. Emergency surgeon-performed hepatobiliary ultrasonography. Br J Surg. 2002 Nov;89(11):1402-4. doi: 10.1046/j.1365-2168.2002.02297.x. PMID 12390381
- [Result] Rozycki GS. Surgeon-performed ultrasound: its use in clinical practice. Ann Surg. 1998 Jul;228(1):16-28. doi: 10.1097/00000658-199807000-00004. PMID 9671062
- [Result] Moore CL, Copel JA. Point-of-care ultrasonography. N Engl J Med. 2011 Feb 24;364(8):749-57. doi: 10.1056/NEJMra0909487. No abstract available. PMID 21345104
- [Result] Allemann F, Cassina P, Rothlin M, Largiader F. Ultrasound scans done by surgeons for patients with acute abdominal pain: a prospective study. Eur J Surg. 1999 Oct;165(10):966-70. doi: 10.1080/110241599750008099. PMID 10574106
- [Result] Lindelius A, Torngren S, Pettersson H, Adami J. Role of surgeon-performed ultrasound on further management of patients with acute abdominal pain: a randomised controlled clinical trial. Emerg Med J. 2009 Aug;26(8):561-6. doi: 10.1136/emj.2008.062067. PMID 19625549
- [Result] Fang R, Pilcher JA, Putnam AT, Smith T, Smith DL. Accuracy of surgeon-performed gallbladder ultrasound. Am J Surg. 1999 Dec;178(6):475-9. doi: 10.1016/s0002-9610(99)00225-1. PMID 10670856
- [Result] Ahmad S, Zafar A, Ahmad M, Ghafoor A, Malik E, Ali A, Qazi UA. Accuracy of surgeon-performed abdominal utrasound for gallstones. J Ayub Med Coll Abbottabad. 2005 Jan-Mar;17(1):70-1. PMID 15929534
- [Result] Shea JA, Berlin JA, Escarce JJ, Clarke JR, Kinosian BP, Cabana MD, Tsai WW, Horangic N, Malet PF, Schwartz JS, et al. Revised estimates of diagnostic test sensitivity and specificity in suspected biliary tract disease. Arch Intern Med. 1994 Nov 28;154(22):2573-81. PMID 7979854
- [Result] Carroll PJ, Gibson D, El-Faedy O, Dunne C, Coffey C, Hannigan A, Walsh SR. Surgeon-performed ultrasound at the bedside for the detection of appendicitis and gallstones: systematic review and meta-analysis. Am J Surg. 2013 Jan;205(1):102-8. doi: 10.1016/j.amjsurg.2012.02.017. Epub 2012 Jun 29. PMID 22748292
- [Result] Lindelius A, Torngren S, Sonden A, Pettersson H, Adami J. Impact of surgeon-performed ultrasound on diagnosis of abdominal pain. Emerg Med J. 2008 Aug;25(8):486-91. doi: 10.1136/emj.2007.052142. PMID 18660395
- [Result] Newcombe RG. Two-sided confidence intervals for the single proportion: comparison of seven methods. Stat Med. 1998 Apr 30;17(8):857-72. doi: 10.1002/(sici)1097-0258(19980430)17:83.0.co;2-e. PMID 9595616
- [Result] Irkorucu O, Reyhan E, Erdem H, Cetinkunar S, Deger KC, Yilmaz C. Accuracy of surgeon-performed gallbladder ultrasound in identification of acute cholecystitis. J Invest Surg. 2013 Apr;26(2):85-8. doi: 10.3109/08941939.2012.697977. Epub 2012 Dec 28. PMID 23273179
- [Result] Scruggs W, Fox JC, Potts B, Zlidenny A, McDonough J, Anderson CL, Larson J, Barajas G, Langdorf MI. Accuracy of ED Bedside Ultrasound for Identification of gallstones: retrospective analysis of 575 studies. West J Emerg Med. 2008 Jan;9(1):1-5. PMID 19561694
- [Result] Shepherd AE, Gogalniceanu P, Kashef E, Purkayastha S, Zacharakis E, Paraskeva PA. Surgeon-performed ultrasound--a call for consensus and standardization. J Surg Educ. 2012 Jan-Feb;69(1):132-3. doi: 10.1016/j.jsurg.2011.09.006. Epub 2011 Nov 3. No abstract available. PMID 22208845
- [Result] Gaspari RJ, Dickman E, Blehar D. Learning curve of bedside ultrasound of the gallbladder. J Emerg Med. 2009 Jul;37(1):51-6. doi: 10.1016/j.jemermed.2007.10.070. Epub 2008 Apr 25. PMID 18439787
- [Derived] Gustafsson C, Lindelius A, Torngren S, Jarnbert-Pettersson H, Sonden A. Surgeon-Performed Ultrasound in Diagnosing Acute Cholecystitis and Appendicitis. World J Surg. 2018 Nov;42(11):3551-3559. doi: 10.1007/s00268-018-4673-z. PMID 29882098
- See also: Statistical procedures — http://OpenEpi.com